CLINICAL TRIAL: NCT00514644
Title: Stroke and Panorama - Analyzing Carotid Endocalcifications
Brief Title: Stroke and Panorama - Analyzing Carotid Endocalcifications (SPACE)
Acronym: SPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Elias Johansson, MD. PhD., Umeå University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EJ-8404
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Carotid Stenoses
Keywords: Panorama; Carotid stenoses
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panorama to Ultrasound (Experimental): 100 asymptotic patients that have findings of calcifications in the area of the carotid arteries when examined with panorama. These persons are examined with carotid ultrasound.
  Interventions: Other: Carotid ultrasound examination
- Ultrasound to Panorama (Experimental): 100 patients with a known carotid stenosis seen on ultrasound will be examined with panorama before any intervention is made. These patients must undergo surgery to be finally included.
  Interventions: Other: Panorama examination

INTERVENTIONS:
Other: Carotid ultrasound examination — Ultrasonographic examination of the carotid arteries to determine the grade of carotid stenosis.
  Arms: Panorama to Ultrasound
Other: Panorama examination — Examination with the odontological radiological method "Panorama", including a frontal verification image
  Arms: Ultrasound to Panorama

SUMMARY:
The odontological radiology method Panorama is known to be able to spot calcifications in the area of the carotid arteries. The calcifications could be carotid stenoses which is affiliated with an increased risk of stroke. The study aims to investigate if panorama examinations can be used as a starting point for further investigation of the carotid arteries.

DETAILED DESCRIPTION:
We intend to examinate 100 consecutive persons that have calcifications in the area of the carotid arteries with carotid duplex-ultrasound. The prevalence of carotid stenoses > 50% (According to the NASCET criteria) in this group is the primary result of interest, answering the most fundamental question - should persons with calcifications in the area of the carotid arteries seen on panorama be screened with ultrasound in order to find asymptomatic carotid stenoses? Since the publication of the ACST and the ACAS studies it is clear that some of these patients might have indications for surgery.

A second part of the study aims to more fully understand what it is that the panorama examination reveals. In this part will 100 patients that are going to undergo surgery to remove their carotid stenoses will be examined with panorama. The carotid plaque that is removed during the surgery will be examined radiologically.

Primary endpoint:

* Subpopulation prevalence of carotid stenoses > 50% in persons with calcifications in the area of the carotid arteries seen in a panoramic examination.

Secondary endpoints:

* Statistical data (sensitivity, specificity, accuracy, likelihood ratio and predictive values) for panorama to find carotid stenoses with ultrasound as gold standard.
* Qualitative description of the relationship between panoramic calcification images and the removed carotid plaques.

AMENDMENT JUNE 2011: The different arms of the study will be published seperately.

ELIGIBILITY:
Inclusion Criteria:

* Panorama to Ultrasound arm:

  * Calcifications in the area of the carotid arteries seen och panorama
* Ultrasound to Panorama arm:

  * Known carotid stenosis > 50%
  * Must undergo carotid endoarterectomy after the panoramic examination

Exclusion Criteria:

* Panorama to Ultrasound arm:

  * Previous cerebrovascular symptoms
  * Below 18 or above 75 years of age
* Ultrasound to Panorama arm:

  * Below 18 or above 90 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2007-08; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The prevalence of carotid stenosis in the group that is examined with carotid ultrasound on the "atheroma on Panoramic examination"-indication

CONTACTS AND LOCATIONS:
Overall Officials: Per G Wester, Prof., Principal Investigator — Umea University; Jan Ahlqvist, Docent, Principal Investigator — Umea University; Eva Levring Jäghagen, Lector, Principal Investigator — Umea University; Elias P Johansson, PhD Student, Principal Investigator — Umea University
Locations (1):
- University Hospital in Umea, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Background] Chambers BR, You RX, Donnan GA. Carotid endarterectomy for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2000;(2):CD001923. doi: 10.1002/14651858.CD001923. PMID 10796451
- [Background] Yin D, Carpenter JP. Cost-effectiveness of screening for asymptomatic carotid stenosis. J Vasc Surg. 1998 Feb;27(2):245-55. doi: 10.1016/s0741-5214(98)70355-6. PMID 9510279
- [Background] Almog DM, Horev T, Illig KA, Green RM, Carter LC. Correlating carotid artery stenosis detected by panoramic radiography with clinically relevant carotid artery stenosis determined by duplex ultrasound. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 Dec;94(6):768-73. doi: 10.1067/moe.2002.128965. PMID 12464905
- [Background] Friedlander AH, Garrett NR, Chin EE, Baker JD. Ultrasonographic confirmation of carotid artery atheromas diagnosed via panoramic radiography. J Am Dent Assoc. 2005 May;136(5):635-40; quiz 682-3. doi: 10.14219/jada.archive.2005.0235. PMID 15966651
- [Result] Johansson EP, Ahlqvist J, Garoff M, Karp K, Jaghagen EL, Wester P. Ultrasound screening for asymptomatic carotid stenosis in subjects with calcifications in the area of the carotid arteries on panoramic radiographs: a cross-sectional study. BMC Cardiovasc Disord. 2011 Jul 13;11:44. doi: 10.1186/1471-2261-11-44. PMID 21752238